CLINICAL TRIAL: NCT04891900
Title: A Single Arm, Multicenter Phase II Clinical Study of TQB2450 (PD-L1 Inhibitor) Plus Anlotinib Combined With Oxaliplatin, Capecitabine in the First-line Treatment of Advanced Gastric Cancer (GC) or Adenocarcinoma of Esophagogastric Junction (AEG)
Brief Title: TQB2450 Plus Anlotinib Combined With Chemotherapy in the Treatment of Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-054-003
Record Dates: First submitted 2021-05-05; First posted 2021-05-19 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; Adenocarcinoma of Esophagogastric Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immune Checkpoint Inhibitors; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 combined with anlotinib, oxaliplatin and capecitabine in the treatment of GC or AEG (Experimental): In this study, all subjects were treated with TQB2450 (PD-L1 inhibitor) plus anlotinib combined with oxaliplatin and capecitabine, once every 3 weeks, six cycles of chemotherapy with oxaliplatin and capecitabine. Subsequently, TQB2450 (PD-L1 inhibitor) combined with anlotinib was maintained until disease progression, intolerable toxicity, withdrawal of informed consent, loss of follow-up or death, or other circumstances that the researcher judged should stop treatment, whichever occurred first.
  Interventions: Drug: TQB2450/Anlotinib hydrochloride/Oxaliplatin/Capecitabine

INTERVENTIONS:
Drug: TQB2450/Anlotinib hydrochloride/Oxaliplatin/Capecitabine — Initial treatment (6 cycles)：
  1. TQB2450：1200 mg , Day 1 ivgtt ,once every 3 weeks
  2. Anlotinib: 10 mg/day orally ，from days 1 to 14 in a 21-day cycle
  3. Oxaliplatin: 130 mg / m2, Day 1 ivgtt ,once every 3 weeks
  4. Capecitabine: 1000 mg / m2, orally, twice a day (once in the morning and once in the evening), from days 1 to 14 in a 21-day cycle Maintenance treatment：
  1）TQB2450: 1200 mg , Day 1 ivgtt , once every 3 weeks 2）Anlotinib: 10 mg/day orally , from days 1 to 14 in a 21-day cycle
  Other Names: PD-L1 inhibitor/Anlotinib

SUMMARY:
This is a prospective one arm phase II clinical study to evaluate the efficacy and safety of TQB2450 (PD-L1 inhibitor), anlotinib combined with oxaliplatin and capecitabine in patients with unresectable locally advanced, recurrent or metastatic gastric cancer or adenocarcinoma of the gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteered to participate in the study and signed the informed consent.
* Age 18-75, both male and female.
* Histology or cytology confirmed HER2/Neu negative (or HER2 / Neu status cannot be determined) non resectable locally advanced or metastatic gastric or esophageal union adenocarcinoma (including signet ring cell carcinoma, mucinous adenocarcinoma and hepatoid adenocarcinoma).
* The time from the end of previous (neoadjuvant) chemotherapy / adjuvant radiotherapy to recurrence was more than 6 months.
* At least one measurable lesion according to RECIST 1.1, which should not be received local treatment such as radiotherapy. If the lesions located in the previous radiotherapy area are confirmed to have progressed and meet the RECIST 1.1 standard, they can also be selected as target lesions.
* ECOG PS 0-1.
* Expected survival ≥ 3 months.
* Adequate organ function as indicated by the following screening laboratory values： Blood test criteria include：

  1. Hemoglobin content (HB) ≥ 90g / L (no blood transfusion within 14 days)
  2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  3. Platelet count (PLT) ≥ 100 × 109/L (no use of IL-11 or TPO within 14 days)
  4. WBC ≥ 4.0 × 109/L (no granulocyte stimulating factor used within 14 days)

Biochemical tests should meet the following standards:

1. Serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN)
2. ALT and AST≤2.5ULN
3. Cr ≤ 1.5 ULN or CCR ≥ 60ml/min, (Cockcroft Gault formula)
4. Serum albumin ≥ 25g/L (2.5g/dL)
5. For patients with liver metastases, AST and ALT must be ≤ 5 x ULN, WBC ≥ 4 × 109 /L, platelets without blood transfusion ≥ 100 × 109 / L, absolute neutrophil count (ANC) ≥ 1.5 × 109 / L, hemoglobin ≥ 90 g / L. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).

Sufficient coagulation function was defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 fold ULN.

* Fertile women were required to take effective contraceptive measures during the study period and at least 180 days after the last administration and chemotherapy.It is suggested that contraceptive measures should be taken at least 3 months before the administration of the study drug; men who are not sterilized must take effective contraceptive measures at least 180 days during the study period, after the last administration and after chemotherapy. It is recommended that contraceptive measures should be taken at least 3 months before the administration of the study drug.
* For example, local treatment of metastatic lesions, such as radiotherapy and ablation, can also be included as long as there are evaluable lesions, and local treatment is not targeted, chemotherapy, immune and other anti-tumor treatment, 28 days after elution.

Exclusion Criteria:

* Allergic to any test drug and its excipients, or with a history of severe allergy, or as a contraindication to the test drug.
* Active or history of autoimmune disease .
* Symptomatic / Asymptomatic brain metastases.
* CT suggests definite ulcerative lesions or stool occult blood positive.
* There was a history of abnormal bleeding one month before admission ( Except epistaxis ).
* Prior allogeneic bone marrow transplantation or organ transplantation
* Congenital pulmonary fibrosis, drug-induced pneumonia, organizing pneumonia, or active pneumonia confirmed by CT.
* HIV positive, active hepatitis B or C, active tuberculosis.
* Uncontrolled cancer pain
* Live attenuated vaccine was injected 4 weeks before the start of the study, or is expected to be injected during the trial or within 5 months after the end of the trial.
* Have received PD-1 / PD-L1 antibody, CTLA-4 antibody, or other treatment for PD-1 / PD-L1 and / or VEGFR inhibitors, or have not recovered from adverse events caused by medication more than 4 weeks ago (i.e., have not recovered to ≤ level 1 or baseline level).
* Systemic application of glucocorticoids or immunosuppressants within 2 weeks before the start of the trial (Note: inhaled glucocorticoids and corticosteroids are allowed).
* Symptomatic central nervous system metastases and / or cancerous meningitis are known. Patients with a history of central nervous system metastasis or spinal cord compression can be enrolled if they have received definite treatment and have stable clinical manifestations 4 weeks after discontinuation of anticonvulsants and steroids before the first administration of the study.
* Hormone contraindications.
* Affect oral medications (e.g. inability to swallow, chronic diarrhea, intestinal obstruction, etc.).
* Peripheral neuropathy ≥ NCI CTCAE 2.
* Uncontrolled or symptomatic hypercalcemia.
* Infections requiring antibiotics within 14 days before the start of the trial.
* Chronic enteritis.
* The load of liver metastasis is more than 50% of the whole liver volume.
* Patients with bone metastases at risk of paraplegia.
* Patients with any severe and / or uncontrolled disease, include:

  1. Patients with poor blood pressure control by antihypertensive drugs (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); patients with grade II or above myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥ 480ms); patients with grade III-IV cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% by NYHA standard.
  2. Active or uncontrolled severe infection.
  3. Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis.
  4. Poor control of diabetes mellitus (FBG > 10mmol / L).
  5. Urine routine examination showed that urine protein was ≥ + +, and 24-hour urine protein was more than 1.0 g.
* Long-term unhealed wounds or fractures.
* Subjects unable to receive peripherally inserted central catheter (PICC) .
* Abnormal coagulation (INR>1.5 or APTT>1.5 ×ULN ), bleeding tendency or thrombolytic or anticoagulant therapy. Known to have inherited or acquired bleeding and thrombotic tendency, such as: hemophilia, blood clotting skills disorder, thrombocytopenia, hypersplenism, etc. Those who had significant coughing up blood 2 months before entering the study, or the daily volume of hemoptysis reached half a teaspoon (2.5 ml) or more. There were significant clinical bleeding symptoms or clear bleeding tendency within 3 months before entering the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer and baseline fecal occult blood ++ And above, or suffering from vasculitis, etc. Long term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥ 300 mg / day or clopidogrel ≥ 75 mg / day).
* Have undergone major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose of the study or expected major surgery during the study treatment period, or non-diagnostic surgery within 4 weeks before the start of the trial.
* A history of gastrointestinal perforation and/or fistula in the 6 months prior to enrollment; or arterial/venous thrombotic events, such as cerebrovascular accidents (except for stable cerebral infarction evaluated by the investigator), deep vein thrombosis, and pulmonary Embolizer.
* Clinically significant pleural and ascites, including any pleural and ascites that can be found on a physical examination, and any pleural and ascites that has been treated in the past or still needs treatment. Only those with a small amount of pleural and ascites on imaging but asymptomatic can be selected if the investigator evaluates that they do not require treatment.
* Suffering from interstitial lung disease that requires steroid therapy.
* Uncontrolled metabolic disorders or other non-malignant tumor organs or systemic diseases or cancer secondary reactions, which can lead to higher medical risks and/or uncertainty in survival evaluation.
* Significantly malnourished patients.
* Have a history of psychotropic drug abuse and can not quit or have mental disorders.
* Have a history of immunodeficiency, including those who have tested positive for HIV or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation.
* History of other primary malignancies, with the exception of the following: 1) Malignant tumors that have completely remitted for at least 2 years before enrollment and no other treatment is required during the study period; 2) Non-melanoma skin cancer or skin cancer that has been adequately treated and has no evidence of disease recurrence Malignant freckle; 3) Carcinoma in situ that has been adequately treated and has no evidence of disease recurrence.
* Pregnant or lactating women.
* According to the judgment of the investigator, those with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.
* Participate in other trials within 30 days before the start of the trial, or plan to participate in other trials while the trial is in progress.
* In case of repetition，enter the group under the most stringent conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | each 2 weeks(Initial treatment) or 3 weeks (maintenance treatment ) up to Progressive Disease（PD） or toxicity intolerable

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | each 2 weeks(Initial treatment) or 3 weeks (maintenance treatment ) up to Progressive Disease（PD） or toxicity intolerable
Duration of Progression-Free Survival (PFS) | each 2 weeks(Initial treatment) or 3 weeks (maintenance treatment ) up to Progressive Disease（PD） or toxicity intolerable
Duration of Overall Survival (OS) | each 2 weeks(Initial treatment) or 3 weeks (maintenance treatment ) up to Progressive Disease（PD） or toxicity intolerable

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Doctor, Principal Investigator — Henan Tumor Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Bie L, Wei C, Luo S, Dong S, Gu Z, Ma Y, Xia Q, Zhang H, Li J, Deng W, Li N. Benmelstobart plus anlotinib and chemotherapy in HER2-negative advanced gastric or gastroesophageal junction adenocarcinoma: A phase 2 study. Cell Rep Med. 2025 Jun 17;6(6):102145. doi: 10.1016/j.xcrm.2025.102145. Epub 2025 May 22. PMID 40409264